CLINICAL TRIAL: NCT03398902
Title: Personalizing Sleep Interventions to Prevent Type 2 Diabetes in Community Dwelling Adults With Pre-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R00NR017416 (NIH); R00NR017416 (NIH)
Record Dates: First submitted 2018-01-05; First posted 2018-01-16 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2023-11

CONDITIONS: PreDiabetes
Keywords: sleep; sleep extension; sleep patterns; type 2 diabetes; glucose regulation; behavioral intervention; adults
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep extension (Experimental): Participants in the sleep extension group will keep daily sleep diaries. Sleep diaries will be reviewed with the participant and an instructor trained in Cognitive Behavioral Therapy for Insomnia (CBTI) on a weekly basis. These weekly sessions will take place by telephone or videoconferencing.
  Interventions: Behavioral: Sleep extension
- Habitual sleep (Active Comparator): Participants in the habitual sleep group will be instructed to keep their habitual bedtimes and wake times. Participants will keep daily sleep diaries that will we reviewed by a study team member each week. These weekly sessions will take place by telephone or videoconferencing.
  Interventions: Other: Habitual sleep

INTERVENTIONS:
Behavioral: Sleep extension — Based on CBTI principles, the instructor will prescribe bed times and wake times each week to allow for gradual increases in sleep opportunity.
  Arms: Sleep extension
Other: Habitual sleep — The study team member will monitor and encourage participants to keep bedtimes and wake times that matched their baseline bedtimes and wake times.
  Arms: Habitual sleep

SUMMARY:
This study will use continuous glucose monitoring and actigraphy to examine whether a personalized, daily sleep extension intervention improves glucose regulation for community dwelling, sleep-restricted adults with pre-diabetes. The randomized controlled trial will include 150 adults with pre-diabetes. Sleep extension and habitual sleep groups will complete daily sleep diaries and participate in a weekly 15-minute telephone call or videoconference meeting with a member of the study team (8 sessions total). Data collection will be at 2 time points: pre-randomization and post-intervention (completion of the 8-week intervention). Changes in the percent time glucose is ≥ 140mg/dL at baseline and post-intervention will be established and compared across the sleep extension and habitual sleep arms.

DETAILED DESCRIPTION:
Diet and exercise interventions have made great strides in preventing and delaying type 2 diabetes (T2D) onset: benefits that surpass pharmacological interventions in some people. Disappointingly, only half the amount of weight loss and wide ranges in T2D risk reduction have been reported when translating these programs into community settings using less intense, more affordable interventions. Low program participation rates, underscored by reports that only 50% of Americans with prediabetes attempt lifestyle modifications, suggest that approaches focused on calorie restriction and physical activity are only effective for select, highly motivated individuals. Expanding success for heretofore resistant groups and optimizing long term maintenance requires novel approaches beyond diet and exercise. One novel approach is improving sleep.

Associations between sleep duration, sleep patterns, and glucose regulation in healthy adults suggest that interventions targeting these dimensions of sleep will improve glucose regulation. Improved insulin sensitivity has been reported in a small community based daily sleep extension study (N= 16), as well as in a 2-day lab based sleep extension study using a personalized "catch up" sleep intervention in healthy adults (N = 19,). Limited by small sample sizes, controlled lab conditions, and the exclusion of persons at greatest risk for T2D, the role of sleep in mitigating T2D risk remains uncertain. Moreover, sleep extension interventions have applied a generic approach to extending sleep despite variability in individual sleep need. The sleep extension intervention in this study will address how to extend sleep based on individual responses to the intervention.

This study will test the effects of a personalized daily sleep extension intervention versus habitual sleep patterns on the percentage of time glucose is 140 mg/dL in sleep restricted community-dwelling adults at high risk for T2D. Wearable sensor technologies (continuous glucose monitoring and accelerometry) will be used. This study will inform person-specific sleep interventions that improve glycemic responses, thus providing treatment for the pre-diabetic state.

Hypothesis: Personalized daily sleep extension will result in a lower % time glucose is ≥ 140 compared to habitual sleep after 8 weeks of treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Glycated hemoglobin (Hemoglobin A1C) greater than or equal to 5.7% and less than 6.5%.
* Restricted sleep defined as less than 6.5 hours average work day sleep (actigraphy confirmed).

Exclusion Criteria:

* type 2 diabetes (Hemoglobin A1C greater than or equal to 6.5%)
* pregnancy or lactation (self-report)
* hemophilia (self-report)
* moderate/severe or severe depression (PHRQ greater than or equal to 15))
* alcohol abuse/dependence (Alcohol Use Disorders Identification Test greater than or equal to 10).
* sleep promoting medications (self-report)
* hypoglycemic agents (except metformin) (self-report)

  --current chemotherapy treatments (self-report)
* Shift work during the past 2 months or planned during intervention period (self-report).
* Trans-meridian travel in the past 4 weeks or planned during intervention period (self-report).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Malone, PhD, Principal Investigator — New York University
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are committed to the principles that NIH has articulated regarding the sharing of study results and resources. The Investigators will make unique research resources readily available for research purposes to individuals within the scientific community after publication. The privacy and rights of participants in the research study will be protected by redacting all identifiers and adopting strategies to minimize the risk of unauthorized disclosure of identifiers in accordance with the data security plan and the participant's Institutional Review Board (IRB)-approved informed consent. The consent language for the R00 study will be worded for possible broad data sharing.
  Sharing Model Organisms Not Applicable Genome Wide Association Studies Not Applicable
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The timeline for submission to an NIH-designated data repository will allow first for publication of findings related to the aims of the R00 study, as well as submission of findings as preliminary data for anticipated grant application(s).
Access Criteria: After data collection is complete, the investigators plan to make the full dataset (redacted of all identifying information) available through the National Sleep Research Resource.
URL: http://www.sleepdata.org

REFERENCES:
- [Background] Cappuccio FP, D'Elia L, Strazzullo P, Miller MA. Quantity and quality of sleep and incidence of type 2 diabetes: a systematic review and meta-analysis. Diabetes Care. 2010 Feb;33(2):414-20. doi: 10.2337/dc09-1124. Epub 2009 Nov 12. PMID 19910503
- [Background] Holliday EG, Magee CA, Kritharides L, Banks E, Attia J. Short sleep duration is associated with risk of future diabetes but not cardiovascular disease: a prospective study and meta-analysis. PLoS One. 2013 Nov 25;8(11):e82305. doi: 10.1371/journal.pone.0082305. eCollection 2013. PMID 24282622
- [Background] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Perreault L, Temprosa M, Mather KJ, Horton E, Kitabchi A, Larkin M, Montez MG, Thayer D, Orchard TJ, Hamman RF, Goldberg RB; Diabetes Prevention Program Research Group. Regression from prediabetes to normal glucose regulation is associated with reduction in cardiovascular risk: results from the Diabetes Prevention Program outcomes study. Diabetes Care. 2014 Sep;37(9):2622-31. doi: 10.2337/dc14-0656. Epub 2014 Jun 26. PMID 24969574
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Schellenberg ES, Dryden DM, Vandermeer B, Ha C, Korownyk C. Lifestyle interventions for patients with and at risk for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Oct 15;159(8):543-51. doi: 10.7326/0003-4819-159-8-201310150-00007. PMID 24126648
- [Background] Yoon U, Kwok LL, Magkidis A. Efficacy of lifestyle interventions in reducing diabetes incidence in patients with impaired glucose tolerance: a systematic review of randomized controlled trials. Metabolism. 2013 Feb;62(2):303-14. doi: 10.1016/j.metabol.2012.07.009. Epub 2012 Sep 7. PMID 22959500
- [Background] Linmans JJ, Spigt MG, Deneer L, Lucas AE, de Bakker M, Gidding LG, Linssen R, Knottnerus JA. Effect of lifestyle intervention for people with diabetes or prediabetes in real-world primary care: propensity score analysis. BMC Fam Pract. 2011 Sep 13;12:95. doi: 10.1186/1471-2296-12-95. PMID 21914190
- [Background] Aziz Z, Absetz P, Oldroyd J, Pronk NP, Oldenburg B. A systematic review of real-world diabetes prevention programs: learnings from the last 15 years. Implement Sci. 2015 Dec 15;10:172. doi: 10.1186/s13012-015-0354-6. PMID 26670418
- [Background] Leproult R, Deliens G, Gilson M, Peigneux P. Beneficial impact of sleep extension on fasting insulin sensitivity in adults with habitual sleep restriction. Sleep. 2015 May 1;38(5):707-15. doi: 10.5665/sleep.4660. PMID 25348128
- [Background] Geiss LS, James C, Gregg EW, Albright A, Williamson DF, Cowie CC. Diabetes risk reduction behaviors among U.S. adults with prediabetes. Am J Prev Med. 2010 Apr;38(4):403-9. doi: 10.1016/j.amepre.2009.12.029. PMID 20307809
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Background] Dunkley AJ, Bodicoat DH, Greaves CJ, Russell C, Yates T, Davies MJ, Khunti K. Diabetes prevention in the real world: effectiveness of pragmatic lifestyle interventions for the prevention of type 2 diabetes and of the impact of adherence to guideline recommendations: a systematic review and meta-analysis. Diabetes Care. 2014 Apr;37(4):922-33. doi: 10.2337/dc13-2195. PMID 24652723
- [Background] Cardona-Morrell M, Rychetnik L, Morrell SL, Espinel PT, Bauman A. Reduction of diabetes risk in routine clinical practice: are physical activity and nutrition interventions feasible and are the outcomes from reference trials replicable? A systematic review and meta-analysis. BMC Public Health. 2010 Oct 29;10:653. doi: 10.1186/1471-2458-10-653. PMID 21029469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community by 1) study flyers, 2) past study participants who agreed to be contacted for future research studies, 3) using Epic to identify and contact potential participants, 4) using research registries such as Research Match, and 5) using a peer recruitment strategy.The first participant enrolled in March 2021 and the last participant enrolled in April 2023.
Pre-assignment Details: Of 393 enrolled participants,191 met inclusion criteria and were randomized to treatment.
Groups:
- Control: Participant received a modified Diabetes Prevention Program Curriculum.
- Sleep Intervention: Participants received a modifed Diabetes Prevention Program curriculum plus a personalized sleep intervention.
Period: Overall Study
Arm/Group | Control | Sleep Intervention
Started | 92 | 99
Completed | 43 | 75
Not Completed | 49 | 24

BASELINE CHARACTERISTICS:
Groups:
- Sleep Intervention: Participants in the sleep extension group will keep daily sleep diaries. Sleep diaries will be reviewed with the participant and an instructor trained in Cognitive Behavioral Therapy for Insomnia (CBTI) on a weekly basis. These weekly sessions will take place by telephone or videoconferencing.
- Control: Participants in the habitual sleep group will be instructed to keep their habitual bedtimes and wake times. Participants will keep daily sleep diaries that will we reviewed by a study team member each week. These weekly sessions will take place by telephone or videoconferencing.
- Total: Total of all reporting groups
Arm/Group | Sleep Intervention | Control | Total
Number analyzed (Participants) | 99 | 92 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.92 (9.03) | 52.80 (8.465) | 52.35 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 58 | 125
  Male | 32 | 34 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 22 | 41
  Not Hispanic or Latino | 79 | 64 | 143
  Unknown or Not Reported | 1 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 12 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 44 | 27 | 71
  White | 40 | 39 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 14 | 19
Percent time Glucose >= 140mg/dL [Mean (Standard Deviation); unit: percentage] — The percent time glucose was >= 140 mg/dL was estimated using continuous glucose monitoring. The average percentage of the time glucose was >= 140mg/dL over the monitoring period was calculated.
  percentage | 5.80 (8.13) | 6.82 (8.57) | 6.29 (8.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Percent Time Glucose is ≥ 140 mg/dL From Pre- to Post-intervention
Description: The primary outcome will be the change in the percent time glucose is ≥ 140mg/dL from pre- to post-intervention estimated from ~7 days of continuous glucose monitoring.
Time Frame: pre-treatment at baseline and post-treatment at ~12 weeks
Measure: Mean (Standard Deviation); unit: Percent time glucose >= 140mg/dL
Groups:
- Control: Participants in the control group will be instructed to keep their habitual bedtimes and wake times. Participants will keep daily sleep diaries that will we reviewed by a study team member each week. These weekly sessions will take place by telephone or videoconferencing.
Arm/Group | Sleep Intervention | Control
Number analyzed (Participants) | 99 | 92
Percent time glucose >= 140mg/dL | 0.38 (4.74) | -0.49 (3.22)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through the 12 week intervention and the following 2-week post-intervention monitoring period.
Groups:
- Sleep Intervention: Participants in the sleep extension group will keep daily sleep diaries. Sleep diaries will be reviewed with the participant and an instructor trained in Cognitive Behavioral Therapy for Insomnia (CBTI) on a weekly basis. These weekly sessions will take place by telephone or videoconferencing.
  Sleep extension: Based on CBTI principles, the instructor will prescribe bed times and wake times each week to allow for gradual increases in sleep opportunity.
- Control: Participants in the habitual sleep group will be instructed to keep their habitual bedtimes and wake times. Participants will keep daily sleep diaries that will we reviewed by a study team member each week. These weekly sessions will take place by telephone or videoconferencing.
  Habitual sleep: The study team member will monitor and encourage participants to keep bedtimes and wake times that matched their baseline bedtimes and wake times.
Arm/Group | Sleep Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/92
Other Adverse Events (participants affected / at risk) | 13/99 | 0/92
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sleep Intervention (N=99) | Control (N=92)
compalints of "not feeling well" (General disorders) | 7 | 0
complaints of a head cold (General disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03398902/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03398902/SAP_001.pdf